CLINICAL TRIAL: NCT06571136
Title: Identification of COVID-19 Infection from Measurement of Exhaled Breath
Brief Title: The Measurement of Chemicals in Exhaled Breath Can Identify If a Person is Infected with COVID-19
Status: Recruiting | Type: Observational
Sponsor: N5 Sensors (Industry)
Collaborators: Providence Health & Services (Other); U.S. Department of Homeland Security (Unknown)
Responsible Party: Sponsor
Other Study IDs: N5-202401; 70RSAT22C00000019 (Other Grant/Funding Number: Department of Homeland Security)
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: Breath testing; COVID-19; Nasal swab
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The type and number of chemicals in exhaled breath are different in people with infection as compared to those without infection. In this study, the breath of people with and without COVID infection will be measured. Changes in the amount and type of chemicals in breath will be used to determine if an individual does or does not have COVID infection. If the measurements of breath are a reliable measure of COVID infection, this device may be used to rapidly screen people who are attending large public events (for example, music concert or baseball game) to minimize the spread of COVID at the event.

DETAILED DESCRIPTION:
N5 Sensors has developed a device that can measure chemical concentrations at parts-per-billion levels (for example, 10 molecules in one-billion molecules is 10 parts-per-billion). This device will be used to measure a variety of chemicals in the exhaled breath of human volunteers. The measured chemicals have been selected based on their presence in the breath of subjects with COVID infection. In addition to measuring breath, samples of mucus from the nose of these same subjects will be collected. These nasal samples will be evaluated to determine the presence of the COVID virus and of COVID infection. Changes in chemicals in the breath will be compared to the presence of COVID or to infection with COVID. This comparison will determine if measurement of breath can be used as a quick and simple measure of COVID infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must complete the consent process
2. Subjects of both sexes must be ≥ 18 and ≤ 70 years old
3. Control subjects must have negative RT-PCR and antigen test
4. COVID subjects must have a positive RT-PCR and/or antigen test.

Exclusion Criteria:

1. Subjects with severe lung disease which would prevent them from providing a breath sample through a large bore tube (e.g., large drinking straw)
2. Subjects with uncontrolled diabetes (e.g., ketoacidosis)
3. Subjects who are routinely exposed to paints, paint thinners, gasoline, varnishes, glues, dry cleaning solvents, or industrial cleaning products
4. Subjects who are daily smokers of cigarettes, e-cigarettes, tobacco products, or marijuana
5. Subjects who have consumed alcohol in the previous 24 hours
6. Have not consumed large amounts of garlic (38 grams) over the prior 24 hours. This amount of garlic can come from approximately 6 garlic cloves or garlic supplement capsules,
7. Subjects who are experiencing respiratory failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who present at a regional emergency department
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-26 (Estimated)

PRIMARY OUTCOMES:
Exhaled chemicals in breath will be compared with COVID status | On the day of enrollment, all measurement will be made over the course of 2 hours.
  Between subjects with and without COVID, changes in the chemical composition of exhaled breath are correlated with markers of COVID infection: 1) antigen testing of nasal mucous sample and 2) RT-PCR testing of nasal mucous sample.
Measurement of chemical composition in exhaled breath | On the day of enrollment, all measurement will be made over the course of 2 hours.
  Each subject will provide two breath samples. Each sample will be analyzed by the RISE device.
Assessment of COVID status using nasal swab. | On the day of enrollment, all measurement will be made over the course of 2 hours.
  Two nasal swabs will be collected for each subject. One nasal swab will be evaluated by antigen testing and the other sample will be analyzed using RT-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Regional Medical Center Everett, Everett, Washington, United States